CLINICAL TRIAL: NCT03880786
Title: Pilot Study: Implantation of a Pudendal PNA Test Lead for Neuromodulation by the ENTRAMI Technique in Case of Chronic Perineal Pain Syndrome.
Brief Title: Implantation of a Pudendal PNA Test Lead for Neuromodulation by the ENTRAMI Technique in Case of Chronic Perineal Pain Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Katleen JOTTARD, Deputy Head of Clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-ENTRAMI
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Pudendal Impingement Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PNE test lead (Experimental)
  Interventions: Device: pudendal PNE test lead

INTERVENTIONS:
Device: pudendal PNE test lead — All patients eligible for release surgery will be implanted a PNE test lead (Medtronic) which will be placed (transforaminal or transgluteally) next to the pudendal nerve, at the level of the ischial spine, after surgical release and connected to an external stimulation device. The PNE lead will be fixed at the ischial-spinal ligament with an absorbable suture to prevent dislocation. If a bilateral dissection is needed, bilateral test leads will be placed. Stimulation will be switched on at the second postoperative day, according to the sensory threshold described by the patient. After three weeks the PNE test lead will be removed at the outpatient clinical visit.

SUMMARY:
Pudendal nerve release surgery in case of pudendal impingement syndrome is well described in literature.Pudendal nerve modulation in case of chronic perineal pain is also a promising technique and some small studies exist. However, in the latter group, patient inclusion criteria are very heterogenous and so conclusions about efficacy are difficult to draw. In the surgery group, outcome results also vary between the different approaches but in general, there is room for improvement. After pudendal nerve release in chronic perineal pain syndrome, it can take up to 6 months before improvement for the patient is recorded. This is partially due to the complex chronic pain syndrome mechanism.

Nothing is known about the possible effect of early neuromodulation at the level of the pudendal nerve after his release.

Recently, two cadaveric studies were published which described a minimal invasive trans gluteal approach for pudendal nerve decompression and a pudendal electrode placement.

In the present trial, the investigators would like to combine the endoscopic trans gluteal pudendal release with pudendal neuromodulation to improve the outcome for patients suffering from pudendal impingement syndrome.

The aim is to improve the results of pain score and quality of life of patients undergoing surgery for pudendal release in case of chronic perineal pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for release surgery
* Patients meeting the five Nantes criteria
* Chronic pain for more than 3 months

Exclusion Criteria:

* Pregnancy
* Progressive neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Maximum Visual Analog Pain scores (VAS) | Change from baseline at first postoperative day
  Linear scale raging from 0 (no pain) to 10 (maximal pain).
Maximum VAS pain scores | Change from baseline at three weeks of stimulation
  Linear scale raging from 0 (no pain) to 10 (maximal pain).
Wexner constipation score | Change from baseline at three weeks of stimulation
  Score computed according to a questionnaire. Score raging form 0 (normal) to 30 (severe constipation)
Fecal incontinence severity index | Change from baseline at three weeks of stimulation
  Score computed according to a questionnaire.Scores range from 0 to 61, where the higher the score, the higher the perceived severity of the fecal incontinence.
Quality of life assessed by the SF-36 questionnaire | Change from baseline at three weeks of stimulation
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. It covers several health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.The recommended scoring system for the SF-36 is a weighted Likert system for each item. The items in the subscales are summed to obtain a summary score for each subscale or dimension. Each of the 8 summary scores is linearly transformed on a scale of 0 (negative to health) to 100 (positive for health).
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-IR ) | Change from baseline at three weeks of stimulation
  The PISQ-IR is a validated evaluation tool which can be used clinically as well as in research for assessment of female sexual function (FSF) in women with female pelvic floor disorders.
Brief Male Sexual Function Inventory (BSFI) | Change from baseline at three weeks of stimulation
  The BSFI questionnaire measures male sexual function.Scores range from 0 (unsatisfactory) to 44 (satisfactory)
Female sexual function index (FSFI) | Change from baseline at three weeks of stimulation
  The FSFI is a brief questionnaire measure of sexual functioning in women. Scores range from 2 (unsatisfactory) to 36 (satisfactory).
Patient Health Questionnaire Mood Scale (PHQ-9) | Change from baseline at three weeks of stimulation
  The purpose of QSP-9 is to gather information on the presence and intensity of depressive symptoms.Scores range from 0 (no depression) to 27 (severe depression).
Score on the DN4 questionnaire | Change from baseline at three weeks of stimulation
  The DN4 (which stands for "Douleur Neuropathique 4") is one of the questionnaires that can be useful in diagnosing neuropathic pain. It ranges from 0 to 10. Values equal to superior to 4 give a diagnostic of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Katleen Jottard, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robert R, Labat JJ, Bensignor M, Glemain P, Deschamps C, Raoul S, Hamel O. Decompression and transposition of the pudendal nerve in pudendal neuralgia: a randomized controlled trial and long-term evaluation. Eur Urol. 2005 Mar;47(3):403-8. doi: 10.1016/j.eururo.2004.09.003. PMID 15716208
- [Background] Possover M. Laparoscopic management of endopelvic etiologies of pudendal pain in 134 consecutive patients. J Urol. 2009 Apr;181(4):1732-6. doi: 10.1016/j.juro.2008.11.096. Epub 2009 Feb 23. PMID 19233408
- [Background] Beco J, Climov D, Bex M. Pudendal nerve decompression in perineology: a case series. BMC Surg. 2004 Oct 30;4:15. doi: 10.1186/1471-2482-4-15. PMID 15516268
- [Background] Heinze K, Hoermann R, Fritsch H, Dermietzel R, van Ophoven A. Comparative pilot study of implantation techniques for pudendal neuromodulation: technical and clinical outcome in first 20 patients with chronic pelvic pain. World J Urol. 2015 Feb;33(2):289-94. doi: 10.1007/s00345-014-1304-7. Epub 2014 Apr 29. PMID 24777254
- [Background] Peters KM, Killinger KA, Jaeger C, Chen C. Pilot Study Exploring Chronic Pudendal Neuromodulation as a Treatment Option for Pain Associated with Pudendal Neuralgia. Low Urin Tract Symptoms. 2015 Sep;7(3):138-42. doi: 10.1111/luts.12066. Epub 2014 Jul 8. PMID 26663728
- [Background] Ploteau S, Robert R, Bruyninx L, Rigaud J, Jottard K. A new endoscopic minimal invasive approach for pudendal nerve and inferior cluneal nerve neurolysis: An anatomical study. Neurourol Urodyn. 2018 Mar;37(3):971-977. doi: 10.1002/nau.23435. Epub 2017 Oct 26. PMID 29072775
- [Background] Jottard K, Bonnet P, Bruyninx L, Ploteau S, De Wachter S. The ENTRAMI technique: Endoscopic transgluteal minimal invasive technique for implantation of a pudendal electrode under full visual control: A cadaver study. Neurourol Urodyn. 2019 Jan;38(1):130-134. doi: 10.1002/nau.23850. Epub 2018 Oct 12. PMID 30311696
- [Derived] Jottard K, Bruyninx L, Bonnet P, Mathieu N, De Wachter S. Pilot study: pudendal neuromodulation combined with pudendal nerve release in case of chronic perineal pain syndrome. The ENTRAMI technique: early results. Int Urogynecol J. 2021 Oct;32(10):2765-2770. doi: 10.1007/s00192-020-04565-1. Epub 2020 Oct 13. PMID 33048179